CLINICAL TRIAL: NCT03552783
Title: Get Your Mind Right: Feasibility of a Mental Health Intervention for African American Fathers in North Omaha
Brief Title: Mental Health Intervention for Black Fathers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0092-18-EP
Record Dates: First submitted 2018-04-16; First posted 2018-06-12 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Mental Health Wellness 1
Keywords: fathers; parenting; African American
MeSH Terms: interventions — Cognitive Behavioral Therapy; Single Person

STUDY DESIGN:
Intervention Model Description: The intervention will be a quasi-experimental study. The participants will be randomized into one of two study arms: Father For a Lifetime (FFL) + Cognitive Behavioral Therapy (CBT) (intervention arm) or FFL only (comparison arm).
Who Masked: Participant
Masking Description: The program coordinator is intimately involved with program participants as his role includes completing the intakes with each participant, implementing the program, and for the purpose of the study, the screening process. To eliminate the bias, the program coordinator will continue to collect intake data and screen the participants. However, we will include a Licensed Mental Health Professional (LIMHP) who will utilize the screening information to complete the comprehensive assessment, randomize, and enroll the participants in the study. In addition, the LIMHP will also complete the follow-up data collection. This will prevent researcher bias during program delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fathers for a Lifetime (FFL) only (Active Comparator): The participants in the comparison arm will receive the standard, 12-week program curriculum of Father For a Lifetime.
  Interventions: Behavioral: Fathers for a Lifetime (FFL) only
- FFL + Cognitive Behavioral Therapy (Experimental): The participants in the intervention will receive will the standard, 12-week program curriculum of Father For a Lifetime and the Cognitive Behavioral Therapy. The intervention will be delivered by a gender and culturally-matched Licensed Mental Health Professional (LIMHP). In addition, the men will receive three one-on-one therapy sessions with a Charles Drew LIMHP that will be completed by the end of the FFL program.
  Interventions: Behavioral: FFL + Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: FFL + Cognitive Behavioral Therapy — Participants in the intervention arm will receive the standard, 12-week program curriculum of Fathers for a Lifetime in addition to 12 weekly, one-hour, group CBT sessions, and three (3), one-hour, one-on-one therapy sessions throughout the 12-week FFL program. We will implement an individual and group CBT mental health intervention that will align with the topics addressed in the FFL weekly curriculum.
  Arms: FFL + Cognitive Behavioral Therapy
Behavioral: Fathers for a Lifetime (FFL) only — The participants in the comparison arm will receive the standard, 12-week program curriculum of Fathers for a Lifetime. The curriculum is broken into three categories:
  1. Personal responsibility
  2. Personal responsibility to your child
  3. Responsibility to your family and community
  Arms: Fathers for a Lifetime (FFL) only

SUMMARY:
The purpose of this study is to examine the feasibility of implementing a mental health intervention, using individual and group Cognitive Behavior Therapy (CBT), embedded into Fathers for a Lifetime; an existing parenting program for fathers. The study will also assess the mental health status and daily functioning of fathers participating in the intervention and comparison arms. The mental health treatments available for parents focused on prevention and treatment of mothers or families but rarely was there a focus on fathers. Our study will use an existing parenting program for fathers to provide a mental health treatment for African American fathers with the intent of creating an effective treatment to screen, diagnosis, increase access to mental health services, and provide mental health treatment. By improving fathers' mental health, we can expect to see improvement in daily functioning, parent-parent interactions, parent-child interactions, increase confidence in parenting skills, and a decrease in parental stress.

DETAILED DESCRIPTION:
The intervention will utilize the Cognitive Behavioral Therapy (CBT), an evidence-based psychotherapeutic approach to addressing mental health issues ranging from anxiety, depression, and other mental illnesses. CBT is based on a cognitive model, the way that individuals perceive a situation is more closely connected to their reaction than the situation itself. The purpose of CBT is to help people focus on how to solve their current problems. The therapist helps the patient learn how to identify distorted or unhelpful thinking patterns, recognize and change inaccurate beliefs, relate to others in more positive ways, and change behaviors accordingly. Participants in the intervention arm will receive 12 weekly, one-hour, group CBT sessions, and three, one-hour, one-on-one therapy sessions throughout the 12-week Father For a LIfetime (FFL) program. We will implement an individual and group CBT mental health intervention that will align with the topics addressed in the FFL weekly curriculum. For instance, the group CBT intervention will examine methods to build resiliency, develop skills to remain calm in stressful situations, learn coping skills when separated from their child/children, and learn how to cope with strained relationships. The FFL curriculum is adapted from the Wise Guys: Male Responsibility Curriculum, an evidence-informed curriculum designed to engage males in the prevention of pregnancies. The curriculum topics are broken into three categories: 1) personal responsibility, 2) responsibility to your child and 3) responsibility to your family and community. Figure 1 below displays the topic description covered each week within each category. The intention of our proposed therapeutic mental health intervention is to improve mental health status utilizing CBT in a group setting and initiating treatment of specific mental illnesses in the one-on-one therapy sessions to meet the unique needs of the father that may not be addressed in a group setting. Participants will receive the intervention immediately after the FFL programming concludes.

The intervention will be delivered by a gender and culturally-matched Licensed Mental Health Professional (LIMHP) who will be trained to deliver the curriculum by the co-investigator and Senior Director of Behavioral Health Services at Charles Drew Health Center. In addition, the men will receive three one-on-one therapy sessions with a Charles Drew LIMHP that will be completed by the end of the FFL program. Participants in the comparison arm will receive the standard, 12-week program curriculum. Our proposed study falls within the T3 translational spectrum, which includes testing an intervention within a community setting by observing and gathering information on implementation to determine feasibility or effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* African American men
* Father
* 19 or older at the time of the enrollment
* Fluent in English (speaking and reading)
* Reside within the specific zip codes: 68104, 68110, 68111, 68112, and 68131

Exclusion Criteria:

* Females
* Not speaking English

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — FFL is open to new, experienced or estranged African American fathers.
Enrollment: 10 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Attrition | 12 weeks post-randomization
  Follow-up rate: participants who completed the 12 weeks program

SECONDARY OUTCOMES:
Mental health status | Baseline; 12 weeks post-randomization
  Defined according to the National Institute of Mental Health definition and DSM-V criteria
Mental health diagnoses | Baseline; 12 weeks post-randomization
  National Institute of Mental Health definition and Diagnostic Statistical Manual (DSM)-V criteria
Daily functioning | Baseline; 12 weeks post-randomization
  Four out of five domains of the Daily Living Activities (DLA-20) Functional Assessment: coping skills, communication, family relationships, and social networking.
Number of FFL participants screened | Baseline
  Number of participants who completed the Intake Form and the DLA-20
Refusal rates for participation | Baseline; 12 weeks post-randomization
  Number of participants who decline to participate in the study
Adherence to study procedures | Baseline; 12 weeks post-randomization
  Participants who successfully followed the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Keyonna M King, DrPH, Principal Investigator — University of Nebraska; Paul Estabrooks, PhD, Study Chair — University of Nebraska
Locations (1):
- Charles Drew Health Center, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Only the entities involved in the study will have access to the participants' data. The data will be collected and temporarily stored at Charles Drew Health Center (the recruitment site). The participants' data will be stored and analyzed at the Center to Reduce Health Disparities/University of Nebraska Medical Center.

REFERENCES:
- [Background] Sinkewicz M, Lee R. Prevalence, Comorbidity, and Course of Depression Among Black Fathers in the United States. Research on Social Work Practice 21(3): 289-297, 2011.
- [Background] Klonoff EA, Landrine H, & Ullman JB. Racial discrimination and psychiatric symptoms among Blacks. Cultural Diversity and Ethnic Minority Psychology 5: 329-339, 1999.
- [Background] Landrine H, Elisabeth A, Klonoff EA. The Schedule of Racist Events: A Measure of Racial Discrimination and a Study of Its Negative Physical and Mental Health Consequences. Journal of Black Psychology 22: 144-168, 1996.
- [Background] Clifford LB, Mavaddat R, Hsu SY. The Experience and Consequences of Perceived Racial Discrimination: A Study of African Americans. Journal of Black Psychology 26: 165-180, 2000.
- [Background] Sellers SL, Bonham V, Neighbors HW, Amell JW. Effects of racial discrimination and health behaviors on mental and physical health of middle-class African American men. Health Educ Behav. 2009 Feb;36(1):31-44. doi: 10.1177/1090198106293526. Epub 2006 Nov 27. PMID 17130248
- [Background] Rosin RD. Perspectives--IJS Issue No. 4, 2009. Int J Surg. 2009 Aug;7(4):277-8. doi: 10.1016/j.ijsu.2009.07.007. Epub 2009 Jul 23. No abstract available. PMID 19631298
- [Background] DeNavas-Walt C, Proctor PD, Smith J. Income, poverty, and health insurance coverage in the United States: 2006. Washington, DC: U.S. Census Bureau. 2007.
- [Background] Huang CC, Warner LA. Relationship characteristics and depression among fathers with newborns. Soc Serv 79: 95-118, 2005.
- [Background] DeKlyen M, Brooks-Gunn J, McLanahan S, Knab J. The mental health of married, cohabiting, and non-coresident parents with infants. Am J Public Health. 2006 Oct;96(10):1836-41. doi: 10.2105/AJPH.2004.049296. Epub 2006 Mar 29. PMID 16571717
- [Background] Amrock SM, Weitzman M. Parental psychological distress and children's mental health: results of a national survey. Acad Pediatr. 2014 Jul-Aug;14(4):375-81. doi: 10.1016/j.acap.2014.02.005. Epub 2014 May 29. PMID 24882378
- [Background] Paulson JF, Dauber S, Leiferman JA. Individual and combined effects of postpartum depression in mothers and fathers on parenting behavior. Pediatrics. 2006 Aug;118(2):659-68. doi: 10.1542/peds.2005-2948. PMID 16882821
- [Background] Kane P, Garber J. The relations among depression in fathers, children's psychopathology, and father-child conflict: a meta-analysis. Clin Psychol Rev. 2004 Jul;24(3):339-60. doi: 10.1016/j.cpr.2004.03.004. PMID 15245835
- [Background] Das Eiden R, Leonard KE. Paternal alcoholism, parental psychopathology, and aggravation with infants. J Subst Abuse. 2000;11(1):17-29. doi: 10.1016/s0899-3289(99)00016-4. PMID 10756511
- [Background] McMahon TJ, Winkel JD, Rounsaville BJ. Drug abuse and responsible fathering: a comparative study of men enrolled in methadone maintenance treatment. Addiction. 2008 Feb;103(2):269-83. doi: 10.1111/j.1360-0443.2007.02075.x. PMID 18199306
- [Background] Beardslee WR, Gladstone TR, Wright EJ, Cooper AB. A family-based approach to the prevention of depressive symptoms in children at risk: evidence of parental and child change. Pediatrics. 2003 Aug;112(2):e119-31. doi: 10.1542/peds.112.2.e119. PMID 12897317
- [Background] Klein DN, Lewinsohn PM, Rohde P, Seeley JR, Olino TM. Psychopathology in the adolescent and young adult offspring of a community sample of mothers and fathers with major depression. Psychol Med. 2005 Mar;35(3):353-65. doi: 10.1017/s0033291704003587. PMID 15841871
- [Background] Lieb R, Isensee B, Hofler M, Pfister H, Wittchen HU. Parental major depression and the risk of depression and other mental disorders in offspring: a prospective-longitudinal community study. Arch Gen Psychiatry. 2002 Apr;59(4):365-74. doi: 10.1001/archpsyc.59.4.365. PMID 11926937
- [Background] Cooke CG, Kelley ML, Fals-Stewart W, Golden J. A comparison of the psychosocial functioning of children with drug-versus alcohol-dependent fathers. Am J Drug Alcohol Abuse. 2004 Nov;30(4):695-710. doi: 10.1081/ada-200037530. PMID 15624545
- [Background] Griffith DM, Neighbors HW, Johnson J. Using national data sets to improve the health and mental health of Black Americans: challenges and opportunities. Cultur Divers Ethnic Minor Psychol. 2009 Jan;15(1):86-95. doi: 10.1037/a0013594. PMID 19209983
- [Background] Yorgason JB, Linville D, Zitzman B. Mental health among college students: do those who need services know about and use them? J Am Coll Health. 2008 Sep-Oct;57(2):173-81. doi: 10.3200/JACH.57.2.173-182. PMID 18809534
- [Background] Nickerson KJ, Helms JE, Terrell F. cultural mistrust, opinions about mental illness, and Black students' attitudes toward seeking psychological help from white counselors. J Counsel Psychol 41: 378-85, 1994.
- [Background] Halgin RP, Weaver DD, Donaldson PE. College students' perceptions of the advantages and disadvantages of obtaining psychotherapy. J of Soc Service Res 8: 75-86, 1986.
- [Background] Hines-Martin V, Malone M, Kim S, Brown-Piper A. Barriers to mental health care access in an African American population. Issues Ment Health Nurs. 2003 Apr-May;24(3):237-56. doi: 10.1080/01612840305281. PMID 12623684
- [Background] Ayalon L, Young MA. Racial group differences in help-seeking behaviors. J Soc Psychol. 2005 Aug;145(4):391-403. doi: 10.3200/SOCP.145.4.391-404. PMID 16050338
- [Background] Barksdale CL, Molock SD. Perceived norms and mental health help seeking among African American college students. J Behav Health Serv Res. 2009 Jul;36(3):285-99. doi: 10.1007/s11414-008-9138-y. Epub 2008 Jul 31. PMID 18668368
- [Background] Bender DS, Skodol AE, Dyck IR, Markowitz JC, Shea MT, Yen S, Sanislow CA, Pinto A, Zanarini MC, McGlashan TH, Gunderson JG, Daversa MT, Grilo CM. Ethnicity and mental health treatment utilization by patients with personality disorders. J Consult Clin Psychol. 2007 Dec;75(6):992-9. doi: 10.1037/0022-006X.75.6.992. PMID 18085915
- [Background] Copeland VC, Butler J. Reconceptualizing access: a cultural competence approach to improving the mental health of African American women. Soc Work Public Health. 2007;23(2-3):35-58. doi: 10.1080/19371910802148263. PMID 19306587
- [Background] Woodward AT, Taylor RJ, Chatters LM. Use of Professional and Informal Support by Black Men with Mental Disorders. Res Soc Work Pract. 2011 Jul;21(3):328-336. doi: 10.1177/1049731510388668. PMID 21686069
- [Background] Douglas County Health Department. Maternal child health (MCH) tables, 2016.
- [Background] McCarter-Spaulding D, Shea S. Effectiveness of Discharge Education on Postpartum Depression. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):168-72. doi: 10.1097/NMC.0000000000000236. PMID 27128643
- [Background] Wozney L, Olthuis J, Lingley-Pottie P, McGrath PJ, Chaplin W, Elgar F, Cheney B, Huguet A, Turner K, Kennedy J. Strongest Families Managing Our Mood (MOM): a randomized controlled trial of a distance intervention for women with postpartum depression. Arch Womens Ment Health. 2017 Aug;20(4):525-537. doi: 10.1007/s00737-017-0732-y. Epub 2017 Jun 7. PMID 28593360
- [Background] Howland M, Armeli S, Feinn R, Tennen H. Daily emotional stress reactivity in emerging adulthood: temporal stability and its predictors. Anxiety Stress Coping. 2017 Mar;30(2):121-132. doi: 10.1080/10615806.2016.1228904. Epub 2016 Oct 1. PMID 27635675
- [Background] Melnyk BM, Feinstein NF, Alpert-Gillis L, Fairbanks E, Crean HF, Sinkin RA, Stone PW, Small L, Tu X, Gross SJ. Reducing premature infants' length of stay and improving parents' mental health outcomes with the Creating Opportunities for Parent Empowerment (COPE) neonatal intensive care unit program: a randomized, controlled trial. Pediatrics. 2006 Nov;118(5):e1414-27. doi: 10.1542/peds.2005-2580. Epub 2006 Oct 16. PMID 17043133
- [Background] Welch MG, Myers MM. Advances in family-based interventions in the neonatal ICU. Curr Opin Pediatr. 2016 Apr;28(2):163-9. doi: 10.1097/MOP.0000000000000322. PMID 26886783
- [Background] Stahl ST, Albert SM, Dew MA, Lockovich MH, Reynolds CF 3rd. Coaching in healthy dietary practices in at-risk older adults: a case of indicated depression prevention. Am J Psychiatry. 2014 May;171(5):499-505. doi: 10.1176/appi.ajp.2013.13101373. PMID 24788282
- [Background] Kuyken W, Hayes R, Barrett B, Byng R, Dalgleish T, Kessler D, Lewis G, Watkins E, Brejcha C, Cardy J, Causley A, Cowderoy S, Evans A, Gradinger F, Kaur S, Lanham P, Morant N, Richards J, Shah P, Sutton H, Vicary R, Weaver A, Wilks J, Williams M, Taylor RS, Byford S. Effectiveness and cost-effectiveness of mindfulness-based cognitive therapy compared with maintenance antidepressant treatment in the prevention of depressive relapse or recurrence (PREVENT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):63-73. doi: 10.1016/S0140-6736(14)62222-4. Epub 2015 Apr 20. PMID 25907157
- [Background] Munshi K, Eisendrath S, Delucchi K. Preliminary long-term follow-up of Mindfulness-based cognitive therapy-induced remission of depression. Mindfulness (N Y). 2013 Dec 1;4(4):354-361. doi: 10.1007/s12671-012-0135-0. PMID 24443660
- [Background] Sandler I, Gunn H, Mazza G, Tein JY, Wolchik S, Berkel C, Jones S, Porter M. Effects of a Program to Promote High Quality Parenting by Divorced and Separated Fathers. Prev Sci. 2018 May;19(4):538-548. doi: 10.1007/s11121-017-0841-x. PMID 28913663
- [Background] Doyle O, Joe S, Caldwell CH. Ethnic differences in mental illness and mental health service use among Black fathers. Am J Public Health. 2012 May;102 Suppl 2(Suppl 2):S222-31. doi: 10.2105/AJPH.2011.300446. Epub 2012 Mar 8. PMID 22401518
- [Background] Demontigny F, Girard ME, Lacharite C, Dubeau D, Devault A. Psychosocial factors associated with paternal postnatal depression. J Affect Disord. 2013 Aug 15;150(1):44-9. doi: 10.1016/j.jad.2013.01.048. Epub 2013 Mar 13. PMID 23489392
- [Background] Waller H, Craig T, Landau S, Fornells-Ambrojo M, Hassanali N, Iredale C, Jolley S, McCrone P, Garety P. The effects of a brief CBT intervention, delivered by frontline mental health staff, to promote recovery in people with psychosis and comorbid anxiety or depression (the GOALS study): study protocol for a randomized controlled trial. Trials. 2014 Jun 27;15:255. doi: 10.1186/1745-6215-15-255. PMID 24973026
- [Background] Sadler P, McLaren S, Klein B, Jenkins M, Harvey J. Cognitive behaviour therapy for older adults experiencing insomnia and depression in a community mental health setting: Study protocol for a randomised controlled trial. Trials. 2015 Nov 27;16:538. doi: 10.1186/s13063-015-1066-6. PMID 26614277
- [Background] Eccleston C, Fisher E, Law E, Bartlett J, Palermo TM. Psychological interventions for parents of children and adolescents with chronic illness. Cochrane Database Syst Rev. 2015 Apr 15;4(4):CD009660. doi: 10.1002/14651858.CD009660.pub3. PMID 25874881
- [Background] Taylor HL, Rybarczyk BD, Nay W, Leszczyszyn D. Effectiveness of a CBT Intervention for Persistent Insomnia and Hypnotic Dependency in an Outpatient Psychiatry Clinic. J Clin Psychol. 2015 Jul;71(7):666-83. doi: 10.1002/jclp.22186. Epub 2015 Apr 23. PMID 25907406
- [Background] Lopez MA, Basco MA. Effectiveness of cognitive behavioral therapy in public mental health: comparison to treatment as usual for treatment-resistant depression. Adm Policy Ment Health. 2015 Jan;42(1):87-98. doi: 10.1007/s10488-014-0546-4. PMID 24692026
- [Background] Beck Institute for Cognitive Behavior Therapy. What is cognitive behavior therapy (CBT)? Retrieved on December 15 from https://beckinstitute.org/get-informed/what-is-cognitive-therapy/.
- [Background] National Institute of Mental Health. RAISE Glossary. Retrieved on December 16, 2017 from https://www.nimh.nih.gov/health/topics/schizophrenia/raise/glossary.shtml.
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Scott RL, Presmanes WS. Reliability and validity of the Daily Living Activities Scale: a functional assessment measure for severe mental disorders. Res Soc Wk Prac 11(3): 373-389, 2001.
- [Background] McGrew JH, Bond GR, Dietzen L, Salyers M. Measuring the fidelity of implementation of a mental health program model. J Consult Clin Psychol. 1994 Aug;62(4):670-8. doi: 10.1037//0022-006x.62.4.670. PMID 7962870
- [Background] Bond GR, Evans L, Salyers MP, Williams J, Kim HW. Measurement of fidelity in psychiatric rehabilitation. Ment Health Serv Res. 2000 Jun;2(2):75-87. doi: 10.1023/a:1010153020697. PMID 11256719
- See also: National Institute of Mental Health. RAISE Glossary. — https://www.nimh.nih.gov/health/topics/schizophrenia/raise/glossary.shtml